CLINICAL TRIAL: NCT04643743
Title: A Retrospective, Observational, Multicentre, Study to Evaluate the Safety and Performance of POLYPATCH ® Vascular Patch
Status: Completed | Type: Observational
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-POL-01
Record Dates: First submitted 2020-11-01; First posted 2020-11-25 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Artery Stenosis, Carotid; Artery Stenosis; Occlusion of Artery; Stroke
Keywords: vascular patch; Polypatch; femoral endarterectomy; carotid endarterectomy; Thrombosis
MeSH Terms: conditions — Carotid Stenosis; Arterial Occlusive Diseases; Stroke; Thrombosis | interventions — Endarterectomy; Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects who did receive POLYPATCH® for vascular angioplasty: Subjects who did receive POLYPATCH® at least one year ago for vascular angioplasty. 2 main sub-populations will be studied depending on location of surgery (carotid and femoral) but data will be collected for all subjects who did receive POLYPATCH.
  Interventions: Device: Endarterectomy

INTERVENTIONS:
Device: Endarterectomy — Endarterectomy is a surgical procedure to remove the atheromatous plaque material, or blockage, in the lining of an artery constricted by the buildup of deposits. It is carried out by separating the plaque from the arterial wall.
  Other Names: Carotid Endarterectomy; Femoral Endarterectomy; Patch Angioplasty

SUMMARY:
POLYPATCH® study is RWE multicentre study which examine short and long-term outcomes of using POLYPATCH® when exposed to a larger and more varied population.

All data will be retrieved from medical charts for each patient from time of surgery (considered as baseline of study) until a maximum of 3 years after surgery.

A minimum of 250 up to a maximum of 300 subjects will be evaluated from 3 to 8 different sites. At least 100 subjects will be evaluated in carotid location and at least 100 in femoral location.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who did receive POLYPATCH® at least one year ago for vascular angioplasty
* Subjects ≥ 18 years old

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will screen all potential subjects and will select those who are appropriate for study inclusion, i.e. adult subjects implanted with POLYPATCH® for at least one year.
  All data will be retrieved from medical charts for each patient from time of surgery (considered as baseline of study) until a maximum of 3 years after surgery.
  A minimum of 250 up to a maximum of 300 subjects will be evaluated from 3 to 8 different sites. At least 100 subjects will be evaluated in carotid location and at least 100 in femoral location.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Change rate of restenosis | within 30 days after surgery and long term (up to 1 year after surgery )
  Measure assessing change target-artery restenosis (defined as 70% or more diameter-reducing stenosis), occlusion, or re-intervention within 1 year after surgery using POLYPATCH®

SECONDARY OUTCOMES:
Procedural success rate | within 30 days after surgery and long term (up to 1 year after surgery )
  * ability to use with no need for using another device,
  * effective vascular closure after endarterectomy procedure,
  * no need to re-operate before patient discharge
target-artery restenosis Target-artery restenosis | within 30 days after surgery and long term (up to 3 years)
  Restenosis can be identified by echo-doppler, CT scan or angiography evaluating the percentage of lumen of vessel but can also be classified as symptomatic vs asymptomatic and/or requiring or not re-intervention.
target-artery re-intervention | within 30 days after surgery and long term (up to 3 years)
  * angioplasty and stenting,
  * surgical bypass,
  * thrombectomy and re-do patchoplasty,
  * evacuation of hematoma.
stroke (ipsilateral and any) | within 30 days after surgery and long term (up to 3 years)
  Stroke is a risk inherent to any surgical intervention, especially vascular surgeries. Although uncommon, stroke in the perioperative period is associated with significant morbidity and mortality in the CEA patient population
transient ischemic attack | 3 years
  within 30 days after surgery and long term (up to 3 years)
myocardial infarction | 3 years
  within 30 days after surgery and long term (up to 3 years)
mortality (cardiovascular and all causes) | within 30 days after surgery and long term (up to 3 years)
  Death is the most dramatic complication one can encounter after vascular procedure. It can result from ipsilateral stroke caused by restenosis or thrombi, patch rupture caused by patch infection, or secondary cardiovascular or neurologic risks caused by the surgery itself
occurrence of other complications | within 30 days after surgery and long term (up to 3 years)
  within 30 days after surgery and long term (up to 3 years)
Operation time | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Armel Plaine, Master, Study Director — Eclevar Medtech
Locations (1):
- Eclevar Medtech, Paris, France